CLINICAL TRIAL: NCT06765057
Title: Effect of Probiotics "Psychobiotics" on Depression in Adults With Pre-Metabolic Syndrome and Metabolic Syndrome in Riyadh City
Brief Title: Effect of Probiotics "Psychobiotics" on Depression and Metabolic Syndrome in Saudi Arabia
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Roaa Ahmed Alkreadees (Other Government)
Responsible Party: Sponsor-Investigator, Roaa Ahmed Alkreadees, Study coordinator and Co-author, King Saud Medical City
Organization: King Saud Medical City (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E-23-7867
Record Dates: First submitted 2024-12-24; First posted 2025-01-09 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Depression Anxiety Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The probiotic and the placebo are packed in plain white sachets, with the study acronym and shelf life printed on them. The sachets are packed in plain white boxes that are all equally labelled with the study title, instructions for use and investigator contact details. Each participant will receive 6 boxes of the same randomization number. The study team will be blinded to the contents of each box. The coordinating investigator of the study team will distribute the numbered boxes to the participants. The investigators have access to the randomization data in case it is necessary to unblind for a serious event. Sealed code break envelopes per participant (located at the investigational site in a restricted-access, fireproof, vault, accessible within 24 hours) will be used and in the event of a code break, the name of the code breaker, the signature, date and time will be recorded on the outside of the envelope. Unblinding will automatically lead to exclusion from the trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Winclove's Ecologic® Barrier Probiotics (Experimental): Patients in the interventional group will consume psychobiotics daily in addition to their antidepressant medication for 12 weeks. All patients will be instructed to take 1 sachet in the morning before breakfast, and 1 sachet at the end of the day before going to bed. The product is a multispecies probiotic formulation consisting of 9 selected probiotic strains by Winclove's Ecologic® Barrier, Amsterdam, The Netherlands. Each participant will receive 6 boxes of the probiotic supplement, each box contains 30 sachets of 3 grams (180 sachets in total). During the period of 12 weeks, each participant will consume 168 sachets. The probiotic supplement is a freeze-dried powder of probiotic mixture at a dose of 2,5 x 109 colony forming units (CFU) per gram. Since participants should consume 2 sachets/day, they will consume 6 grams in total which equals 1.5 × 10^10 CFU.
  Interventions: Dietary Supplement: Winclove's Ecologic® Barrier Probiotics
- Control (Placebo Comparator): Patients in the control group will consume similar sachets that are identical in physical appearance. The placebo is composed of the carrier of the probiotic product, that is maize starch and maltodextrins but contains no bacteria.
  Interventions: Dietary Supplement: Winclove's Ecologic® Barrier Probiotics Placebo

INTERVENTIONS:
Dietary Supplement: Winclove's Ecologic® Barrier Probiotics — The investigational product is a multispecies probiotic formulation consisting of 9 selected probiotic strains: the following bacterial strains: Bifidobacterium bifidum W23, Bifidobacterium lactis W52, Lactobacillus acidophilus W37, Lactobacillus brevis W63, Lactobacillus casei W56, Lactobacillus salivarius W24, Lactococcus lactis W19 and Lactococcus lactis W58.
  Arms: Winclove's Ecologic® Barrier Probiotics
Dietary Supplement: Winclove's Ecologic® Barrier Probiotics Placebo — The placebo is composed of the carrier of the probiotic product that are identical in physical appearance, it includes maize starch and maltodextrins but contains no bacteria.
  Arms: Control

SUMMARY:
The goal of this clinical trial is to assess the effect of commercial multi-strains psychobiotics supplementation as an ad-on therapy on depressive symptoms and metabolic syndrome components (HDL-C, FPG, TGs, WC, BP) in adult depressed patients with pre-metabolic syndrome and metabolic syndrome. The second goal is to explore the effect of commercial multi-strains psychobiotics supplementation on the anthropometric measurement (weight, body mass index (BMI)) in adult depressed patients with pre-metabolic syndrome and metabolic syndrome. The main questions they aim to answer are:

* Will commercial multi-strains psychobiotics supplementation help to ease depressive symptoms as an ad-on therapy in patients with pre-metabolic syndrome and metabolic syndrome?
* Will commercial multi-strains psychobiotics supplementation improve anthropometric measurements and metabolic syndrome components (WC, FPG, BP, TGs, HDL-C) in depressed patients? Researchers will compare psychobiotics to a placebo (a look-alike substance that contains no drug) to see if psychobiotics work to improve depression and metabolic syndrome components.

Participants will:

* Be examined for depression, anxiety, and metabolic syndrome components (waist circumference, diabetes, blood pressure, triglycerides, and high-density lipoprotein).
* Be asked to conduct laboratory tests to determine the inclusion and exclusion criteria.
* Be given probiotics/ placebo to consume every day for 3 months (12 weeks).
* Repeat the examination and laboratory tests to determine the results.
* Be followed up weekly for adverse events and to insure their compliance with the study instructions.
* Be followed up after 4 weeks as an end-visit and will conduct the examination and the laboratory blood tests.

DETAILED DESCRIPTION:
Recently, the United Nations (UN) announced depression as the leading cause of disability worldwide. According to the World Health Organization (WHO), depression can increase the risk of suicide and death. Its prevalence increased globally since 2005 from 4.4% and reached 18.4% in 2015 accounting for about 322 million of the population. Based on the study of the Global Burden of Disease (GBD) from 195 countries around the world including Saudi Arabia, depression incidence increased from 172.27 million to 258.16 million from 1990 to 2017 most of whom is from major depressive disorder (MDD).

In addition, according to the Saudi National Mental Health Survey in 2016, 34% of Saudis were having psychiatric disorders and 80% of those with severe situations did not attempt any health care. Moreover, the prevalence of MDD among Saudis was 0.6% and it was one of the top-rated mental health cases in Saudi Arabia. Not only that but also, a cross-sectional study showed that the incidence of depression increased even more among Saudis during the pandemic of coronavirus disease-19 (COVID-19) to be 20.9%.

Depression is characterized by a persistent feeling of sadness, loss of interest, feeling of low self-esteem, loss of energy, decreased or increased appetite, trouble sleeping, and thoughts of suicide. Basically, depression is categorized into two main categories which are MDD and persistent depressive disorder (known as dysthymia). Depression can impair the quality of life and well-being. Unfortunately, it can also affect health negatively by causing comorbid diseases such as cancer, heart disease, inflammation, and neurological and metabolic disorders.

According to Al-Khatib et al (2022), one of the metabolic disorders associated with depression is metabolic syndrome (MetS). The International Diabetes Federation (IDF) defined the MetS as the occurrence of three or more symptoms of the following: central obesity with waist circumference (WC) for men ≥ 94 centimeters while for women ≥ 80 centimeters, increased fasting plasma glucose (FPG) ≥ 100 mg/dl, increased blood pressure (BP) to ≥ 130 /≥ 85 mmHg, increased triglycerides (TGs) to equal or above 150 mg/dl, reduced high-density lipoprotein cholesterol (HDL-C) for men to < 40 mg/dl while for women < 50 mg/dl. Yin et al., 2013 defined the pre-metabolic syndrome (Pre-MetS) as the occurrence of at least two components of MetS that do not reach the diagnostic of MetS. As a matter of fact, depression can lead to MetS and vice versa. About 30% of individuals with depression have MetS; meanwhile, about 41% of individuals with depression and MetS also have high levels of inflammation. Individuals with inflammation tend to have obesity and MetS. Thus, in 2007, it was proposed that the onset of depression with comorbid MetS is called "MetS type II" in which a combination of neuronal, psychological, and metabolic disorder happens. Furthermore, Gawlik-Kotelnicka and Strzelecki mentioned in their recent review the term "metabolic depression" to depict the relationship between depression, obesity, and MetS.

Recently, it has been suggested that gut microbiota modulation by a combination of probiotics and anti-depressant is an effective treatment. Since the bidirectional relationship between brain and gut health was confirmed, the accumulated body of evidence revealed that mental health is impacted by what is called the gut-brain axis (GBA) in which the gut microbiome can affect brain health through special microorganisms known as psychobiotics. Psychobiotics are special types of probiotics; they are specified to positively influence neurotransmitters, endocrinal hormones, and anti-inflammatory cytokines. They are a supporting therapy as an add-on therapy for mood disorders and depression with little or no side effects. To our knowledge, there are no clinical trials conducting in Saudi Arabia to investigate the impact of probiotics efficiency on depressive symptoms, anthropometric measurement, and MetS components in adult patients which is the aim of this experimental study.

ELIGIBILITY:
Inclusion Criteria:

* Major Depression Disorder (MDD) patients on antidepressants for at least 4 weeks or more.
* MDD patients with pre-metabolic syndrome (at least 2 of the MetS components) and metabolic syndrome (at least 3 of the following components: central obesity with WC for men ≥ 94 centimeters while for women ≥ 80 centimeter, increased FPG ≥ 100 mg/dl, increased BP to ≥ 130 / ≥ 85 mmHg, increased TGs equal or above 150 mg / dl, increased HDL cholesterol for men to < 40 mg / dl while for women < 50 mg / dl) (IDF., 2006).
* MDD patients with other comorbid diseases such as anxiety.

Exclusion Criteria:

* Patients using any other supplements to improve mood.
* Patients using pre/pro/symbiotics supplement or antibiotics during the last 3 weeks before the intervention.
* Patients with chronic diseases (cardiac, renal, or hepatic diseases)
* Patients with gastro intestinal diseases (Crohn's disease, ulcerative colitis).
* Patients with infectious diseases (HIV/AIDS).
* Cancer patients or those undergoing chemotherapy.
* Patients with food allergies such as gluten intolerance or lactose intolerance.
* Pregnant and breastfeeding women.
* Patients with modified antidepressant dose during interventional period or receiving psychotherapy during the intervention.
* Patients with thyroid disorder.
* Patients following a diet to lose weight during the intervention.
* Diabetic patients who are insulin-dependent.
* patients receiving injections or medications to lose weight (Ozempic, Mounjaro …etc) either 3 weeks before or during the intervention.
* Patients using plasma-lipid lowering drug for less than 1 month before the intervention.
* Patients with substance abuse including alcohol addiction.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-02 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Psychological Assessment (depression1) | at baseline, after the end of the 12th week of the intervention, and after 4 weeks post-intervention follow-up (end visit).
  • Depression will be diagnosed clinically using the validated Arabic translated Patient Health Questionary 9 (PHQ-9) in Saudi population to assess the severity of depression as a self-report scale for patients in both groups. The minimum score is 0 while the maximum score is 27; the higher the score the more severe the depression is. Scores 0-4 means no depression; scores 5-9 means mild depression; scores 10-14 means moderate depression; score 15-19 means moderately severe, and 20-27 means severe depression.
Psychological Assessment (depression2) | at baseline, after the end of the 12th week of the intervention, and after 4 weeks post-intervention follow-up (end visit).
  • Hamilton Depression Rating Scale (HDRS) will be also used as a clinician-rated scale to evaluate the severity of depression symptoms. The most commonly used versions in are either a 17- or a 21-item scale, but this study uses the 21-item scale. The scoring of the severity of the depressive symptoms is based on 17 items. It is scored between 0 (not present) and 4 (severe) points using either a three-point or a five-point scale and summed up to obtain the total score. Scores 0-7 represent the absence or remission of depression; scores between 8-16 represent mild depression; scores between 17-23 represent moderate depression, and scores equal to 24 and above represent severe depression.
Psychological Assessment (Anxiety) | at baseline, after the end of the 12th week of the intervention, and after 4 weeks post-intervention follow-up (end visit).
  • Generalized Anxiety Disorder-7 (GAD-7) scale will be added to assess anxiety. Each of the 7 items is scored from 0 to 3, the GAD-7 scale score ranges from 0 to 21; the higher the score the more severe the anxiety is. Scores 0-4 means no anxiety; scores 5-9 means mild anxiety; scores 10-14 means moderate anxiety; score 15-21 means severe anxiety.
Anthropometric Measurements | at baseline, after the end of the 12th week of the intervention, and after 4 weeks post-intervention follow-up (end visit).
  Height and weight will be combined to calculate the body mass index (BMI). BMI will be measured through dividing individual's weight in kilograms by height in square meter. Lower than 18.5 means underweight; 18.5 to lower than or equal 25 means normal weight; 25.0 to lower than or equal 30 means overweight; 30.0 or above means obese (Centers for Disease Control and Prevention (CDC), 2020).
Metabolic Syndrome Components (Waist circumference) | at baseline, after the end of the 12th week of the intervention, and after 4 weeks post-intervention follow-up (end visit).
  Central obesity will be measured through waist circumference (WC) by placing non-stretchable meter around the waist above the bone of the hip equally; the tape should be tightened lightly without pressure on skin (Whitney & Rolfes, 2020). WC for men is ≥ 94 centimeters while for women ≥ 80 centimeters (Alberti, Zimmet, & Shaw, 2006).
Metabolic Syndrome Components (Medical Assessments/ Laboratory Tests) | at baseline, after the end of the 12th week of the intervention, and after 4 weeks post-intervention follow-up (end visit).
  Blood samples will be collected out on venous blood after fasting for 12 h. Blood samples in each visit will be collected in 3 tubes and the value will be 3 ml in each tube.
  i. Fasting Plasma Glucose: pre-diabetic is more than 100 mg/dl to 125 mg/dl (Alberti, Zimmet, & Shaw, 2006).
  ii. Hemoglobin A1C (HgA1C): pre-diabetic HbA1c is between 5.7 - 6.5% (Alberti, Zimmet, & Shaw, 2006).
  iii. Triglycerides: more than 150 mg/dl (Alberti, Zimmet, & Shaw, 2006). iv. High Density Lipoprotein-Cholesterol: less than 40 mg/dl in men and less than 50 mg/dl in women (Alberti, Zimmet, & Shaw, 2006).
Metabolic Syndrome Components (Medical Assessments/ Blood Pressure) | at baseline, after the end of the 12th week of the intervention, and after 4 weeks post-intervention follow-up (end visit).
  • Blood pressure for both groups will be measured three times sequentially at 1-min interval using the standardized method, the average between the three readings will be used as study variable (if more than 130 mmHg systolic BP/or more than 85 mmHg diastolic BP).

CONTACTS AND LOCATIONS:
Locations (1):
- King Saud University Medical City, Riyadh, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with the probiotics company (Winclove's). KSUMC will provide Winclove with "raw data" a complete overview of the final results of the study after analysis and after anonymization to comply with applicable regulations, but not with patient identifying data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Until January 15th, 2027.
Access Criteria: Through electronic files.

REFERENCES:
- [Background] Altwaijri YA, Al-Habeeb A, Al-Subaie AS, Bilal L, Al-Desouki M, Shahab MK, Hyder S, Sampson NA, King AJ, Kessler RC. Twelve-month prevalence and severity of mental disorders in the Saudi National Mental Health Survey. Int J Methods Psychiatr Res. 2020 Sep;29(3):e1831. doi: 10.1002/mpr.1831. Epub 2020 Aug 15. PMID 33245602
- [Background] Al-Khatib Y, Akhtar MA, Kanawati MA, Mucheke R, Mahfouz M, Al-Nufoury M. Depression and Metabolic Syndrome: A Narrative Review. Cureus. 2022 Feb 12;14(2):e22153. doi: 10.7759/cureus.22153. eCollection 2022 Feb. PMID 35308733
- [Background] AlHadi AN, Alarabi MA, AlMansoor KM. Mental health and its association with coping strategies and intolerance of uncertainty during the COVID-19 pandemic among the general population in Saudi Arabia: cross-sectional study. BMC Psychiatry. 2021 Jul 28;21(1):382. doi: 10.1186/s12888-021-03370-4. PMID 34320930
- [Background] Gawlik-Kotelnicka O, Strzelecki D. Probiotics as a Treatment for "Metabolic Depression"? A Rationale for Future Studies. Pharmaceuticals (Basel). 2021 Apr 20;14(4):384. doi: 10.3390/ph14040384. PMID 33924064
- [Background] Gold SM, Kohler-Forsberg O, Moss-Morris R, Mehnert A, Miranda JJ, Bullinger M, Steptoe A, Whooley MA, Otte C. Comorbid depression in medical diseases. Nat Rev Dis Primers. 2020 Aug 20;6(1):69. doi: 10.1038/s41572-020-0200-2. PMID 32820163
- [Background] Alberti KG, Zimmet P, Shaw J. Metabolic syndrome--a new world-wide definition. A Consensus Statement from the International Diabetes Federation. Diabet Med. 2006 May;23(5):469-80. doi: 10.1111/j.1464-5491.2006.01858.x. PMID 16681555
- [Background] Liu Q, He H, Yang J, Feng X, Zhao F, Lyu J. Changes in the global burden of depression from 1990 to 2017: Findings from the Global Burden of Disease study. J Psychiatr Res. 2020 Jul;126:134-140. doi: 10.1016/j.jpsychires.2019.08.002. Epub 2019 Aug 10. PMID 31439359
- [Background] Park C, Brietzke E, Rosenblat JD, Musial N, Zuckerman H, Ragguett RM, Pan Z, Rong C, Fus D, McIntyre RS. Probiotics for the treatment of depressive symptoms: An anti-inflammatory mechanism? Brain Behav Immun. 2018 Oct;73:115-124. doi: 10.1016/j.bbi.2018.07.006. Epub 2018 Jul 18. PMID 30009996
- [Background] Sharma R, Gupta D, Mehrotra R, Mago P. Psychobiotics: The Next-Generation Probiotics for the Brain. Curr Microbiol. 2021 Feb;78(2):449-463. doi: 10.1007/s00284-020-02289-5. Epub 2021 Jan 4. PMID 33394083
- [Background] Vlainic JV, Suran J, Vlainic T, Vukorep AL. Probiotics as an Adjuvant Therapy in Major Depressive Disorder. Curr Neuropharmacol. 2016;14(8):952-958. doi: 10.2174/1570159x14666160526120928. PMID 27226112
- See also: Major Depressive Disorder — http://www.ncbi.nlm.nih.gov/books/NBK559078/
- See also: UN health agency reports depression now 'leading cause of disability worldwide' — https://news.un.org/en/story/2017/02/552062
- See also: Depression and Other Common Mental Disorders: Global Health Estimates — http://www.who.int/publications-detail-redirect/depression-global-health-estimates
- See also: Apolipoprotein B/apolipoprotein A1 ratio is a good predictive marker of metabolic syndrome and pre-metabolic syndrome in Chinese adolescent women with polycystic ovary syndrome — http://pubmed.ncbi.nlm.nih.gov/22672648/